CLINICAL TRIAL: NCT01944605
Title: Intestinal Ischemia as a Stimulus for Systemic Inflammatory Response After Cardiac Arrest
Acronym: TICA
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: HM15326
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Cardiac Arrest; Reperfusion Injury
Keywords: Endotoxin; Cytokine; Metabolism
MeSH Terms: conditions — Heart Arrest; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma Blood serum Whole blood Stool Expired Gas
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Arrest patients undergoing Therapeutic Hypothermia: Cardiac Arrest subjects with Return Of Spontaneous Circulation (ROSC) and undergoing treatment with Therapeutic Hypothermia will undergo sampling of blood, stool, and expired gas data at physiologically predetermined time points.

SUMMARY:
Out-of-hospital cardiac arrest (CA) is a leading public health problem causing nearly one third of a million deaths annually in the US, accounting for half of all cardiovascular deaths and surpassing deaths from stroke, heart failure, and breast and lung cancer combined. Twenty to fifty percent of CA patients (pts) can be resuscitated initially but many die before hospital discharge or suffer permanent neurologic damage. Therapeutic hypothermia (TH) improves survival and neurological outcomes. Despite aggressive, targeted post arrest management, including TH, approximately 50% of pts die before leaving the hospital due to global ischemia-reperfusion injury (IRI) known as the "post arrest syndrome", 1 which is a sepsis-like state characterized by elevated markers of cellular inflammation and injury. It is believed that TH works by decreasing the body's basal metabolic rate (BMR) and attenuating the systemic inflammatory response (SIR). However, specific triggers of the intense pro-inflammatory response are unclear. This "gap" in knowledge must be closed to identify targeted therapy to decrease IRI and improve outcomes.

Blood flow to the gut is decreased markedly and intestinal tissue becomes ischemic during CA and CPR, particularly when vasoconstrictor drugs such as epinephrine, are given. IRI of the intestine increases intestinal permeability leading to intestinal microbial translocation and endotoxin release that can stimulate and perpetuate systemic inflammation and cause subsequent multi-organ dysfunction. Endotoxin also increases body temperature and energy expenditure and may attenuate TH induced reductions in BMR and hence, decrease efficacy. The purpose of this novel pilot study is to detect systemic endotoxin release following CA in humans and determine association with cytokine activation, and BMR alterations during TH.

DETAILED DESCRIPTION:
Hypothesis 1 Intestinal ischemia during and following Caridac Arrest leads to increased gut permeability and endotoxin release that stimulates the Systemic Inflammatory Response that is responsible for subsequent death and disability after resuscitation.

Hypothesis 2: Different degrees of systemic endotoxin activity variably affect Basic Metabolic Rate during Therapeutic Hypothermia

Serial samples of blood, stool and expired gas will be measured at predetermined timepoints after ROSC from cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

Adult, Cardiac Arrest with ROSC receiving Therapeutic Hypothermia-

Exclusion Criteria:

* Age < 18
* Cardiac Arrest of traumatic etiology
* Known to be pregnant
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients resuscitated from Cardiac Arrest successfully and undergoing therapeutic hypothermia will be evaluated for potential inclusion
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03-30 (Actual); Study Completion 2014-03-30 (Actual)

PRIMARY OUTCOMES:
Detection of Endotoxin Activity | 48 hours
  Endotoxin activity will be measured by the Endotoxin Activity Assay and values . of >0.4 EA units will be used as the "cut-off" for the presence of pathological endotoxin.

SECONDARY OUTCOMES:
Detection of sCD14 | 48 hours
  To demonstrate activation of endotoxin by the immune system and "upstream" physiologic changes necessary for systemic endotoxemia to occur
Detection of stool lactoferrin and stool α1-antitrypsin | 48 hours
  To demonstrate evidence of intestinal inflammation and permeability that can lead to endotoxemia and "downstream" cellular inflammatory responses responsible for end organ damage
Detection and quantification of inflammatory cytokines | 48 hours
  To demonstrate an association with the primary outcome
BMR measurement elevation | 48 hours
  To determine its association with endotoxemia and cytokine. BMR is being measured to determine if pts with higher levels of endotoxin and cytokines have higher BMR and therefore blunted therapeutic value of TH

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Peberdy, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States